CLINICAL TRIAL: NCT01822340
Title: A Phase II, Randomized, Active Controlled, Open Label Study of Safety and Efficacy of HM10560A a Long-acting rhGH-HMC001 Conjugate in Treatment of Subjects Suffering From Adult Growth Hormone Deficiency (AGHD)
Brief Title: Safety and Efficacy Study of Recombinant Human Growth Hormone in Adult Growth Hormone Deficiency Patients
Acronym: HM10560A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-HM10560A-201
Record Dates: First submitted 2013-03-25; First posted 2013-04-02 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Adult Growth Hormone Deficiency
Keywords: AGHD
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 (Experimental): Once weekly HM10560A
  Interventions: Drug: HM10560A
- Cohort 2 (Experimental): Once weekly HM10560A
  Interventions: Drug: HM10560A
- Cohort 3 (Experimental): Once weekly HM10560A
  Interventions: Drug: HM10560A
- Cohort 4 (Experimental): Biweekly HM10560A
  Interventions: Drug: HM10560A
- Cohort 5 (Active Comparator): Once daily Genotropin
  Interventions: Drug: Genotropin

INTERVENTIONS:
Drug: HM10560A — Once weekly HM10560A
  Other Names: LAPS-rhGH
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4
Drug: Genotropin — Once daily Genotropin
  Other Names: Genotropin 5.3mg
  Arms: Cohort 5

SUMMARY:
The purpose of this study is to assess the safety, tolerability and Pharmacokinetic/ Pharmacodynamic (PK/PD) profile of three doses of HM10560A on an every week (EW) regime and one dose on every other week (EOW) regime administered for a period of 24 weeks initial study.

DETAILED DESCRIPTION:
* To select the optimal dose and dosing regimen of HM10560A for the subsequent phase III study on the basis of the safety and PK/PD profile after 24 weeks of treatment
* To assess the long term safety of HM10560A when administered in optimal dose range and dose frequency for additional 48 weeks (followed with 2 weeks safety follow up)

ELIGIBILITY:
Inclusion Criteria:

* GHDA subjects, males and females, of age between 23 and 60 years as defined in the Consensus Guidelines for the Diagnosis and Treatment of Adults with GH Deficiency II (2007) as well as American Association of Clinical Endocrinologists Medical Guidelines for Clinical Practice for Growth Hormone Use in Growth Hormone-Deficient Adults and Transition Patients (2009);
* r-hGHdrug naïve or any registered or investigational r-hGH replacement therapy was not given for more than 6 months before the screening.
* Body Mass Index (BMI, kg/m2) of both male and female patients must be between 22.0 to 35.0 kg/m2.
* Female patients must have a negative serum pregnancy test at inclusion.
* Confirmed to be negative for anti r-hGH antibodies at the time of screening.
* Willing and able to provide written informed consent prior to performing any study procedures.

Exclusion Criteria:

* Patients with childhood onset of GHD treated with r-hGH before the age of 18.
* Current antitumor therapy.
* Subjects presenting with any clinically significant ECG abnormality.
* Evidence of intracranial hypertension.
* Significant hepatic dysfunction (persistent elevation of alanine transaminase [ALT] or aspartate transaminase [AST] >1.5 x upper limit of normal).
* Pregnancy and breastfeeding;

Ages: 23 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2011-10; Primary Completion 2015-06 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change of IGF-I levels in function of time, and dose strengths | baseline, 1,2,3,4,5,6,7,8,9,10,11,12,13,14,15,16,17,18 months
  The results from each month minus baseline

SECONDARY OUTCOMES:
IGF-I SDS; changes to baseline in IGF-I SDS | baseline, 1,2,3,4,5,6,7,8,9,10,11,12,13,14,15,16,17,18 months
  The results from each month minus baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Hanmi Pharmaceutical, Budapest, Hungary